CLINICAL TRIAL: NCT05614687
Title: Art as Healing: A Community-informed Art-based Programme (CiAbP) for Reintegrating Ex-offenders Into Society in Nigeria
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teesside University (Other)
Responsible Party: Principal Investigator, Tarela Ike, Dr, Teesside University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0000-0003-0516-0313b
Record Dates: First submitted 2022-11-05; First posted 2022-11-14 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Trauma; Depression; Anxiety and Fear
Keywords: Trauma; Anxiety and Fear
MeSH Terms: conditions — Wounds and Injuries; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community-informed art-based programme (CiAbP) (Experimental): The CiAbP sessions will cover relevant aspects of art, such as poetry, spoken words, painting, drawing, literature, and music, in tackling trauma and negative attitudes towards ex-offenders reintegration.
  Interventions: Behavioral: Community-informed art-based programme
- Government intervention involving media messages (Active Comparator): It will involve media messages from the National Orientation Agency devoid of CiAbP and other media sources on materials such as health and public awareness.
  Interventions: Other: Government Media Intervention

INTERVENTIONS:
Behavioral: Community-informed art-based programme — The Community-informed art-based programme is an intervention incorporating art in the form of for example poetry and drawings in addressing trauma and encouraging community attitudes towards the positive reintegration of ex-offenders.
  Arms: Community-informed art-based programme (CiAbP)
Other: Government Media Intervention — Government Media Intervention involving media content from the National Orientation Agency and other media sources
  Arms: Government intervention involving media messages

SUMMARY:
The goal of this pilot experimental study is to test a community-informed art-based programme in improving community members trauma from crime and to aid the reintegration of ex-offenders into society.

The main question it aims to answer are:

• What is the feasibility in terms of recruitment, retention, adherence to the intervention and communities/victims' satisfaction with CiAbP to promote healing and improve the successful reintegration of ex-offenders into society?

Participants will be randomly allocated into two groups. The first group, the intervention group, will receive the Community-informed Art-based programme (CiAbP). The second group will receive government intervention involving media messages from the National Orientation Agency devoid of CiAbP. The CiAbP. sessions will cover relevant aspects of art, such as photo story, story telling, poetry, and drawing in tackling trauma and negative attitudes towards ex-offenders reintegration.

Researchers will compare CiAbP group with the media orientation group to see if there are differences between a change in attitude towards ex-offenders' reintegration at base line, end of intervention and three months follow up.

ELIGIBILITY:
Inclusion Criteria:

* Community members with previous experience of trauma
* Aged 18+ years and are residents in areas including Lagos/Delta states and its environs.
* Able to give informed consent,
* Speak the English language,
* Able to partake in baseline, pre-, post- and three-month follow-up data collection.

Exclusion Criteria:

* The exclusion criteria are those not meeting the study's inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Trauma Screening Questionnaire | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in traumatic experience is being assessed
  Change in traumatic experience is being assessed Change in traumatic experience is being assessed
Belief in Redeemability Scale v2 | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in of attitude towards ex-offenders' reintegration is being assessed
Service Satisfaction Scale | Change is being assessed at baseline, at 12 weeks end of intervention, at 3-months post-intervention
  Change in service satisfaction is being assessed

CONTACTS AND LOCATIONS:
Overall Officials: Tarela Ike, Dr, Principal Investigator — Teesside University

IPD SHARING:
Plan to Share IPD: No